CLINICAL TRIAL: NCT00948740
Title: Phase III Study of the Effect of Vitamin D Repletion on Urinary Calcium Excretion in Kidney Stone Formers With Vitamin D Deficiency and High Urinary Calcium
Brief Title: The Effect of Vitamin D on Urinary Calcium Excretion in Kidney Stone Formers With High Urinary Calcium
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jie Tang, MD,M.Sc, Jie Tang, M.D., M.Sc., Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009P000533
Record Dates: First submitted 2009-07-27; First posted 2009-07-29 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Vitamin D Deficiency; Nephrolithiasis
Keywords: vitamin D
MeSH Terms: conditions — Vitamin D Deficiency; Nephrolithiasis | interventions — Ergocalciferols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ergocalciferol (Experimental): After signing informed consent, all participants who meet the study criteria will receive ergocalciferol 50,000 IU weekly for 8 weeks. After completing the ergocalciferol course, participants will take a maintenance dose of cholecalciferol 1,000 IU daily.
  Interventions: Drug: vitamin D (ergocalciferol)

INTERVENTIONS:
Drug: vitamin D (ergocalciferol) — The intervention is oral ergocalciferol 50,000 IU per week for 8 weeks
  Other Names: ergocalciferol

SUMMARY:
The investigators hypothesize that a 3 month course of vitamin D supplementation to treat 25(OH)D deficiency in stone formers with high levels of 24-hour urinary calcium will not increase urinary calcium excretion by greater than 10%.

DETAILED DESCRIPTION:
We plan to conduct a clinic-based interventional study of 30 patients followed at Brigham and Women's Hospital with history of nephrolithiasis, urinary calcium excretion between 200 and 400 mg/day, and 25-vitamin D deficiency (defined as serum level ≤ 25ng/ml). The intervention is oral ergocalciferol 50,000 IU per week for 8 weeks [1], and each participant will serve as his own control. The outcome is the change in urinary calcium excretion. The planned study duration is 3 months. We will have greater than 95% power to detect a 10% increase in 24-hour urinary calcium

ELIGIBILITY:
Inclusion Criteria:

* History of nephrolithiasis
* 25(OH)D deficiency (defined as serum level ≤ 25ng/ml) within 3 months of enrollment
* 24-hour urinary calcium excretion > 199 mg/day and < 400 mg/day (measured less than 6 months prior to study enrollment)

Exclusion Criteria:

* Non-Caucasian
* Women of child-bearing age (age < 50)
* Known uric acid, cystine, or struvite stone disease
* Hypercalcemia (serum calcium > 10.4 mg/dl within the past 12 months)
* Gross hematuria within the past 6 months
* Acute stone event within the past 2 months
* Recent stone intervention within the past 1 month
* Suspected or known secondary causes of hypercalciuria such as primary hyperparathyroidism, sarcoidosis, hyperthyroidism, or malignancy (except non-melanoma skin cancer)
* Addition or dose change of medicines potentially affecting urinary calcium since enrollment 24-hour urine collection (including diuretics, magnesium supplements, potassium supplements, potassium citrate, and vitamin D supplementation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-08; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Urinary calcium level after treatment with ergocalciferol will be compared with the pre-treatment level. The primary outcome is the change in urinary calcium excretion. | 1-2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jie Tang, M.D., M.Sc, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States